CLINICAL TRIAL: NCT06625983
Title: Colorectal Cancer Screening Decision Support Tool in the Primary Care Bundle Questionnaire
Brief Title: Use of a Colorectal Cancer Screening Decision Support Tool in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen J. Blumenthal, MD, MPH, Internist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024P000687
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer Control and Prevention; Colorectal Cancer Screening; Shared Decision Making; Decision Aid
Keywords: colorectal cancer screening; shared decision making; electronic health record; randomized controlled trial; decision tool
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Practices will be randomized to receive the decision tool or not receive the decision tool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CRC decision tool (Experimental): intervention arm
  Interventions: Other: CRC decision tool
- control (No Intervention): control arm

INTERVENTIONS:
Other: CRC decision tool — CRC decision tool included in the primary care bundle questionnaire
  Other Names: intervention
  Arms: CRC decision tool

SUMMARY:
The research question we pose is, Does a colorectal cancer (CRC) screening decision support tool offered in advance of primary care visits increase CRC screening completion rates? Our work aims to answer this question by evaluating the effectiveness of an MGB decision support tool to 1) promote informed decisions about CRC screening for average risk patients ages 45-75, 2) deploy a decision support tool as part of a primary care bundle questionnaire, and 3) support patients in completing their preferred method of CRC screening.

DETAILED DESCRIPTION:
As part of usual care, a CRC screening electronic decision support tool developed by Mass General Brigham has been integrated into Epic. This decision support tool is part of routine clinical care and is sent electronically to patients aged 45-75 who receive the Annual Visit Primary Care Screening Bundled Questionnaire in advance of their annual visit. Patients complete the tool on Patient Gateway prior to the visit or via an iPad at the visit. The decision support tool guides patients through the CRC screening options (e.g., FIT, colonoscopy, Cologuard) to help them select their preferred screening method. As part of routine care, the patient will be prompted to complete the tool as part of the bundled questionnaire, and the results will be available in the Epic encounter in the Screenings tab with the other screening bundle responses. The primary care clinician can then discuss the options and/or screening preference with the patient. Depending on what the patient and clinician decide, a CRC screening test may be ordered for the patient. As a secondary outcome, a random sample of 1000 patients will be surveyed to understand their involvement in the decision making process and 300 providers will be surveyed to understand how the decision tool impacted the conversation with the patient. The IRB to conduct surveys of patients and providers was approved by the Mass General Brigham IRB (Protocol # 2024P002568).

ELIGIBILITY:
Inclusion Criteria:

Adults aged 45-75 overdue for CRC screening at average risk of CRC have an annual visit scheduled with participating practices

Exclusion Criteria:

* high risk of CRC

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80000 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
CRC screening completion | 12 months
  Assessment of electronic health record data to determine completion of CRC screening by any modality

SECONDARY OUTCOMES:
Provider Experience | During the 6 month intervention phase
  Provider-reported question: Did you feel the CRC screening tool informed or affected your conversations in any way?
Shared Decision Making Process Measure | During the 6 month intervention phase
  Patient-reported survey question about involvement in the decision making process.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Blumenthal, MD, Principal Investigator — Massachusetts General Hospital; Karen Sepucha, PhD, Study Director — MGH
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified data will be made available upon request
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The IPD will be available once the study is completed and after approval by the IRB.
Access Criteria: Requests will be reviewed by the PI and the IRB.